CLINICAL TRIAL: NCT01232725
Title: Clinical Epidemiologic and Biologic Studies of Donor Human Milk and Breastfeeding
Brief Title: Donor Human Milk and Neurodevelopmental Outcomes in Very Low Birthweight (VLBW) Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarah T Colaizy (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Tarah T Colaizy, Associate Professor of Pediatrics, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200708746; K23HD057232 (NIH)
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Neurodevelopmental Outcomes of VLBW Infants
Keywords: BSID III; Human Milk; Donor Human Milk; Preterm infant; Breastfeeding
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donor Human Milk (Experimental): VLBW infants randomized to be fed donor human milk, fortified as appropriate, for all feedings for which maternal milk is not available, including infants who receive no maternal milk
  Interventions: Dietary Supplement: Donor Human Milk
- Preterm Formula (Experimental): VLBW infants randomized to receive preterm infant formula for any feedings for which maternal milk is unavailable, including infants receiving no maternal milk
  Interventions: Dietary Supplement: Donor Human Milk

INTERVENTIONS:
Dietary Supplement: Donor Human Milk — Donor Human Milk, obtained from the Mother's Milk of Iowa, a HMBANA milk bank

SUMMARY:
Breastfeeding is an important health-promoting behavior. Human milk is the ideal diet for all infants, optimizes intellect, and provides protection against infectious and atopic diseases in childhood as well as decreasing risks for obesity, hypertension and other chronic diseases. Infants with the highest risk of life-long disability, very low birthweight (VLBW) preterm infants, are breastfed at some of the lowest rates in the US. Maternal milk is not always available, and pasteurized donor human milk is an alternative that requires investigation. Whether donor milk conveys health and developmental advantages similar to those bestowed by maternal milk is unknown. By determining the effects of donor milk on health and developmental outcomes when compared to preterm infant formula, the investigators seek to optimize outcomes in this fragile population. The hypothesis of our donor milk research is that a donor human milk diet in non-maternal milk fed VLBW infants is associated with better neurodevelopmental outcome scores at 18-22 months adjusted age than a preterm infant formula diet.

ELIGIBILITY:
Inclusion Criteria:

* <1501 g weight at birth

Exclusion Criteria:

* chromosomal anomalies
* congenital heart disease
* congenital disorders known to impair neurodevelopment

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2009-08; Primary Completion 2014-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Cognitive scale score of the Bayley Scales of Infant Development, III | 18 - 22 months' adjusted age
  We will administer the BSID III to all subjects at 18-22 mo of age, adjusted for prematurity. We will compare the scores between subjects who received donor human milk to those who received preterm infant formula

SECONDARY OUTCOMES:
Late Onset sepsis | 4 months
  We will compare rates of in-hospital confirmed late onset sepsis in VLBW infants receiving donor human milk and preterm formula
length of hospital stay | 4 months
  We will compare the length of initial hospital stay between infants who receive donor human milk and those who receive preterm infant formula

CONTACTS AND LOCATIONS:
Overall Officials: Tarah T Colaizy, MD, MPH, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact PI to discuss data sharing

REFERENCES:
- [Derived] Quigley M, Embleton ND, Meader N, McGuire W. Donor human milk for preventing necrotising enterocolitis in very preterm or very low-birthweight infants. Cochrane Database Syst Rev. 2024 Sep 6;9(9):CD002971. doi: 10.1002/14651858.CD002971.pub6. PMID 39239939